CLINICAL TRIAL: NCT03905148
Title: A Phase 1b, Open-Label, Dose-escalation and Expansion Study to Investigate the Safety, Pharmacokinetics and Antitumor Activities of a RAF Dimer Inhibitor BGB-283 in Combination With MEK Inhibitor PD-0325901 in Patients With Advanced or Refractory Solid Tumors
Brief Title: Study of the Safety and Pharmacokinetics of BGB-283 (Lifirafenib) and PD-0325901 (Mirdametinib) in Participants With Advanced or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Collaborators: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-283/PD-0325901-AU-001
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — BGB-283; mirdametinib

STUDY DESIGN:
Intervention Model Description: Part A will consist of dose escalation and dose-finding components to establish the max tolerated dose and/or recommended Phase 2 dose Part B will investigate efficacy and further evaluate the PK, safety, and tolerability of the combination of PD-0325901 and BGB-283 (lifirafenib).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A: Dose Escalation/Dose finding Dose Level Cohorts ranging in dose levels and dose regimens. (Experimental): Combination doses of, Mirdametinib at once a day and lifirafenib at once a day And Mirdametinib at twice a day and lifirafenib at once a day
  Interventions: Drug: Lifirafenib; Drug: mirdametinib
- Part B: Expansion (Experimental): Approximately 20 participants with NRAS mutated solid tumors will be enrolled
  Interventions: Drug: Lifirafenib; Drug: mirdametinib

INTERVENTIONS:
Drug: Lifirafenib — RAF Dimer Inhibitor
  Other Names: BGB-283
Drug: mirdametinib — MEK Inhibitor
  Other Names: PD-0325901

SUMMARY:
This is a 2-part Phase 1b study of BGB-283 (lifirafenib) and PD-0325901 (mirdametinib) combination in participants with tumors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Able to provide informed consent
2. Age 18 on day of signing informed consent form (ICF) or of the legal age of consent in the jurisdiction in which the study is taking place
3. Advanced or metastatic, unresectable tumors (other than patients with tumors of the brain or central nervous system) who have experienced disease progression

   * Part A: NSCLC, CRC, ovarian cancer, endometrial cancer, thyroid cancer, melanoma, pancreatic cancer, and other)
   * Part B: NRAS mutated solid tumors must have a known mutation status and a histologically or cytologically confirmed advanced or refractory solid tumor. Up to 40% Melanoma and Up to 20% CRC.
4. Must have archival tumor tissue or agree to tumor biopsy
5. Measurable disease per RECIST 1.1
6. Eastern Cooperative Oncology Group performance status of less than or equal to 1
7. Life expectancy is greater than 12 weeks of the signing of ICF.
8. Adequate organ function and no transfusion within 14 days of first dose.
9. Females are of non-child bearing potential or willing to use contraception.
10. Males vasectomized or agree to use contraception.

Key Exclusion Criteria:

1. Central Nervous System metastasis
2. Any retinal pathology considered to be a risk factor for central serous retinopathy
3. History of glaucoma
4. Active parathyroid disorder or history of malignancy associated hypercalcemia
5. Clinically significant cardiac disease within the past 6 months of signing ICF.
6. LVEF less than 50%
7. Abnormal QT interval at Screening
8. Severe uncontrolled systemic disease
9. HIV
10. Clinically significant active or known history of liver disease. (Hepatitis B and Hepatitis C)
11. Hemorrhage or bleeding event at NCI-CTCAE v5.0 Grade 3 or higher within 28 days of first dose.
12. history of or ongoing Von Willebrand disease and/or other past or present bleeding disorders
13. Increased serum calcium
14. Inability to swallow oral medications
15. Ongoing radiation therapy or radio-cytotoxic therapy within prior 4 weeks. No chemotherapy, immunotherapy, biologic therapy, hormonal, or molecular targeted therapy within prior 2 weeks
16. Concomitant systemic or glucocorticoid therapy within 2 weeks
17. Major surgical procedure or significant traumatic injury within 4 weeks prior to first dose or anticipates need for major surgery while on study
18. Concomitant medicines that are strong CYP3A inhibitors
19. History of toxicity from another RAF, MEK, ERK inhibitor requiring discontinuation of treatment from these drugs
20. Underlying medical conditions in investigator's opinion to be unfavorable to be a part of the study
21. Has been administered a live vaccine within 4 weeks (28 days) of initiation of study treatment. NOTE: injectable seasonal vaccines for influenza and COVID-19 are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and are not allowed.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Adverse Events and Serious Adverse Events | Approximately 2 years from date of the participants enrollment
  Incidence and severity of AEs and SAEs and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
The incidence of DLT events and treatment-emergent AEs (TEAEs) | Approximately 2 years from date of the participants enrollment
Objective response rate based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 in participants with selected tumor types | Approximately 2 years from date of the participants enrollment

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - University of California Los Angeles, Santa Monica, California
  - MD Anderson, Houston, Texas
- Australia (4):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - The Prince of Wales Private Hospital - Specialist Medical Randwick, Randwick, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Desai J, Gan H, Barrow C, Jameson M, Atkinson V, Haydon A, Millward M, Begbie S, Brown M, Markman B, Patterson W, Hill A, Horvath L, Nagrial A, Richardson G, Jackson C, Friedlander M, Parente P, Tran B, Wang L, Chen Y, Tang Z, Huang W, Wu J, Zeng D, Luo L, Solomon B. Phase I, Open-Label, Dose-Escalation/Dose-Expansion Study of Lifirafenib (BGB-283), an RAF Family Kinase Inhibitor, in Patients With Solid Tumors. J Clin Oncol. 2020 Jul 1;38(19):2140-2150. doi: 10.1200/JCO.19.02654. Epub 2020 Mar 17. PMID 32182156